CLINICAL TRIAL: NCT03052881
Title: Robotic Retinal Dissection Device Trial
Acronym: R2D2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16/LO/005
Record Dates: First submitted 2017-01-04; First posted 2017-02-14 (Actual); Last update posted 2020-06-18 (Actual); Status verified 2020-02

CONDITIONS: Epiretinal Membrane; Retinal Hemorrhage
MeSH Terms: conditions — Epiretinal Membrane; Retinal Hemorrhage | interventions — Robotic Surgical Procedures

STUDY DESIGN:
Intervention Model Description: Parallel assignment
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Robot assisted surgery (Experimental): To investigate use of an intraocular robotic system to assist the surgeon in performing one of two operation: i) epiretinal, or inner limiting, membrane peel and ii) displacement of sub macular haemorrhage.
  Interventions: Device: Robot assisted surgery
- Control (No Intervention): A control group of patients underwent either i) epiretinal, or inner limiting, membrane peel and ii) displacement of sub macular haemorrhage without the use of a robot i.e. the surgery was done in the standard manner.

INTERVENTIONS:
Device: Robot assisted surgery — The PRECEYES Surgical System is a robotically assistive device developed by PRECEYES Medical Robotics, a Dutch-based research group at the Technische Universiteit Eindhoven. It has been designed to enhance surgical precision, specifically for vitreoretinal eye surgery. The device provides accuracy beyond human capabilities of <10μm in all directions (x, y, z planes). The surgeon is always in control of the instrument by manipulating the motion controller.
  Arms: Robot assisted surgery

SUMMARY:
The purpose of the study is to determine whether use of a robotic system improves the precision and therefore safety of high precision steps in retinal surgery. Two common surgical scenarios (ERM/ILM peel and sub retinal haemorrhage displacement surgery) that require a high degree of precision to avoid damage to the retina have been chosen for this trial. These steps also have been selected because they allow a clearly definable outcome measure e.g. time taken to complete a specific step in the operation. The main issue here is that the patients will be undergoing this procedure regardless of enrolment in the trial - the only difference being that for study participants the surgeon will perform parts of the operation with the assistance of the robot.

DETAILED DESCRIPTION:
This trial will be a prospective interventional surgical case series to pilot the use of a robotic device in retinal surgery. Specifically, the investigators will determine whether particular operations are performed more quickly and safely with robotic assistance. The PRECEYES Surgical System is a robotically assistive device developed by PRECEYES Medical Robotics, a Dutch-based research group at the Technische Universiteit Eindhoven. It has been designed to enhance surgical precision, specifically for vitreoretinal eye surgery. The device provides accuracy beyond human capabilities of <10μm in all directions (x, y, z planes). The surgeon is always in control of the instrument by manipulating the motion controller. Patients undergoing one of two operations will be invited to enroll in the study (i.e. consent for the following operations is an eligibility criteria for the study itself): i) those undergoing epiretinal or inner limiting membrane peel, ii) those undergoing subretinal haemorrhage displacement surgery. The study will involve the surgeon performing specific surgical steps of these operations, that require very high levels of precision, with the assistance of the robot. Efficiency, accuracy and safety data will be collected. Eligible study participants will be recruited from the cohort of patients attending the outpatient clinics of the Oxford Eye Hospital who require either ERM/ILM peel or sub retinal haemorrhage displacement surgery. The expected duration and frequency of pre- and post-operative follow up will be identical to standard NHS care for these particular operations i.e. no additional study visits or procedures will be required.

ELIGIBILITY:
Inclusion Criteria:

1. Participant is willing and able to give informed consent for i) participation in the trial ii) for the surgery itself e.g. standard NHS consent form.
2. Males or females aged 18 - 90 years.
3. Standard vitreoretinal operation deemed necessary by the ophthalmologist, specifically: injection of subretinal tissue plasminogen activator for treatment of sub retinal haemorrhage, or peeling of epiretinal and/or inner limiting membrane.
4. Patients must be deemed fit for surgery.
5. In the Investigator's opinion, the participant is able and willing to comply with all trial requirements.
6. Willing to allow his or her General Practitioner or Consultant, to be notified of participation in the trial (not required for the control arm).

Exclusion Criteria:

-

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2019-07-23 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
Intra-operative retinal micro-trauma | 3 months
  To explore the safety of the PRECEYES surgical robot assisted surgeon in two specific eye surgery procedures during steps that require the greatest manual precision. A count of the number of iatrogenic retinal micro-haemorrhages and/or inadvertent instrument touches of the retina will be made. This outcome measure will be assessed at the time of surgery and followed post-operatively using optical coherence tomography scans of the macula.

SECONDARY OUTCOMES:
Duration of robotic assisted surgery compared to standard surgery | Intra-operative i.e. 1 day.
  To investigate the speed of the PRECEYES surgical robot assisted surgeon in initiating membrane removal from the retina compared with the standard of care (manual) technique. The duration of steps performed with the assistance of the robot will be compared to the standard operative technique.
Accuracy of instrument positioning in the subretinal space during subretinal injection, measured by visualising the cannula tip position with an integrated optical coherence tomography (OCT) operating microscope. | Intra-operative i.e. 1 day.
  To investigate the accuracy of the PRECEYES surgical robot assisted surgeon in performing subretinal injection of tissue plasminogen activator (tPA). The cannula tip position will be documented using real-time OCT. Where possible, a comparison to the standard technique will be performed. Deviation in an x, y or z plane from the desired optimal position in the subretinal space will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Robert E MaLaren, DPhil FRCOphth, Principal Investigator — University of Oxford
Locations (1):
- University of Oxford, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Anonymised data may be shared with other researchers as per Study Protocol and Research Participant Consent form.

REFERENCES:
- [Derived] Cehajic-Kapetanovic J, Xue K, Edwards TL, Meenink TC, Beelen MJ, Naus GJ, de Smet MD, MacLaren RE. First-in-Human Robot-Assisted Subretinal Drug Delivery Under Local Anesthesia. Am J Ophthalmol. 2022 May;237:104-113. doi: 10.1016/j.ajo.2021.11.011. Epub 2021 Nov 14. PMID 34788592
- See also: A video of the device can be viewed at this website — http://www.preceyes.nl